CLINICAL TRIAL: NCT02534883
Title: Cervical Ripening in Postmenopausal Women: A Randomized, Double Blind, Placebo Controlled Trial
Brief Title: Cervical Ripening in Postmenopausal Women
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not able to meet enrollment
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Donald Gregory Ward, M.D., MD, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 25065
Record Dates: First submitted 2015-08-25; First posted 2015-08-28 (Estimated); Results first posted 2018-07-12 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-06

CONDITIONS: Stenosis of Cervix
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): Group 1 will received 200ug of misoprostol, to be placed into the posterior vaginal fornix 12 hours and 2 hours before their scheduled surgery (a total of 400ug of misoprostol).
  Interventions: Drug: Misoprostol
- Group 2 (Placebo Comparator): Group 2 will received placebo (empty gelatin capsule), to be placed into the posterior vaginal fornix 12 hours and 2 hours before their scheduled surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Misoprostol — To be place vaginally
  Other Names: Cytotec
  Arms: Group 1
Drug: Placebo — To be placed vaginally
  Other Names: non active drug
  Arms: Group 2

SUMMARY:
Misoprostol (Cytotec) 200ug vaginally will be given to patients 12 hours and 2 hours pre-operatively (before surgery) for a total of 400ug to ripen, soften or relax the cervix for dilation (opening). This is to assist with the insertion of a hysteroscope (the surgical instrument) into the uterus for all operative hysteroscopic procedures requiring dilation above 5 mm.

Time required for cervical dilatation will be recorded. Start time will be when the smallest dilator is placed into the endocervical canal, and stop time recorded when the desired cervical dilation is achieved with the largest dilator. Depending on the procedure, desired dilation may range between 5-10mm. Time will serve as a surrogate for operative ease of dilatation.

The investigators will compare the two groups in terms of medication, resistance, dilation time and size, side effects and surgical complications.

DETAILED DESCRIPTION:
This study will be a randomized, double blinded, placebo controlled trial.

Patients will be assigned by chance to receive 200ug of misoprostol or placebo (empty gelatin capsule) vaginally twice (for a total of 400ug). There is no standard of care, but to receive misoprostol or not are both accepted practices and that Standard of Care is for the clinicians to use clinical judgment .

Patients will be randomized to one of the following treatment regimens:

Group 1 will received 200ug of misoprostol, to be placed into the posterior vaginal fornix 12 hours and 2 hours before their scheduled surgery (a total of 400ug of misoprostol). St. Mary's pharmacy will prepare capsules with each containing 200ug of misoprostol.

Group 2 will received placebo (empty gelatin capsule), to be placed into the posterior vaginal fornix 12 hours and 2 hours before their scheduled surgery.

The two groups, will be compared in terms of side effects, resistance, dilation time, size and surgical complication.

Randomization will occur using a computer program called Research Randomizer, http://www.randomizer.org/form.htm. A set of 100 non-unique numbers will be randomized. Once the randomization list is generated, envelopes will be made. Based on the randomizer results a folder slip of paper with the treatment (misoprostol or placebo) written on it will be placed in sequential numbered envelopes. The number on the envelope will be the patients code number. An unblinded member of the research team will open the randomized envelope, and log into a master drug log the randomization.

The medication and/or placebo will be place in numbered sequentially bottles with a master drug log containing which is misoprostol and which is placebo. Each bottle will have child proof lids for dispensing and will be labeled misoprostol 200ug/each/placebo), physician name (Ward) and contact number, and "For investigational use only" will also be noted.

The unblinded staff will notify the research member consenting the patient and inform them of what number bottle to give to the patient, in the office before surgery

ELIGIBILITY:
Inclusion Criteria:

* 45-80yrs of age
* Postmenopausal (amenorrhea for greater than 1 year)
* May or may not be using hormone replacement therapy
* Scheduled or to be scheduled for hysteroscopy/resectoscopy procedures

Exclusion Criteria:

* Pregnant
* Known Cancer
* Known hypersensitivity to prostaglandins.
* Those who are breastfeeding

Ages: 45 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Ward, MD, Principal Investigator — St. Louis University
Locations (1):
- St. Mary's Health Center, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Misoprostol Group: Group 1 will receive 200 ug of misoprostol to be placed into the posterior vaginal fornix 12 hours and 2 hours before the scheduled surgery (a total of 400 ug misoprostol).
  Misoprostol: To be placed vaginally
- Placebo Group: Group 1 will receive placebo (empty gelatin capsule) to be placed into the posterior vaginal fornix 12 hours and 2 hours before the scheduled surgery.
  Placebo: To be placed vaginally
Period: Overall Study
Arm/Group | Misoprostol Group | Placebo Group
Started | 8 | 3
Completed | 0 | 0
Not Completed | 8 | 3
Not completed — Early Termination | 8 | 3

BASELINE CHARACTERISTICS:
Population: Data not compiled because of early termination
Groups:
- Misoprostol Group: Group 1 will receive 200 ug of misoprostol to be placed into the posterior vaginal fornix 12 hours and 2 hours before the scheduled surgery (a total of 400 ug misoprostol).
  Misoprostol: To be placed vaginally
  Baseline characteristics not compiled because of early termination.
- Placebo Group: Group 1 will receive placebo (empty gelatin capsule) to be placed into the posterior vaginal fornix 12 hours and 2 hours before the scheduled surgery.
  Placebo: To be placed vaginally
  Baseline characteristics not compiled because of early termination.
- Total: Total of all reporting groups
Arm/Group | Misoprostol Group | Placebo Group | Total
Number analyzed (Participants) | 8 | 3 | 11
Age, Categorical [Count of Participants; unit: Participants] — Population: 11 enrolled. One participant withdrew because her surgery was cancelled and not rescheduled.
  Data sheet completed at time of surgery and thus only available for 10 participants.
  Participants
    number analyzed (Participants) | 7 | 3 | 10
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 4 | 2 | 6
    >=65 years | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 11 enrolled. One participant withdrew because her surgery was cancelled and not rescheduled.
  Data sheet completed at time of surgery and thus only available for 10 participants.
  years
    number analyzed (Participants) | 7 | 3 | 10
    (all) | 62.3 (5.2) | 58.7 (6.1) | 61.2 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 11
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Efficacy (Cervical Ripening)
Description: To evaluate the efficacy of two doses of 200ug of misoprostol (for a total of 400ug), administered vaginally, on cervical ripening before diagnostic and operative hysteroscopic procedures in postmenopausal women (amenorrhea greater than 1 year). Efficacy is represented by time to dilation.
Time Frame: At time of surgery/cervical dilation
Population: Outcome measures presented below.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 7 | 3
minutes | 1.9 (1.1) | 1.4 (.4)

2. Secondary Outcome: Number of Recorded Side Effects.
Description: Secondary aim: to evaluate if cervical ripening with misoprostol reduces side effects
Time Frame: At time of surgery/cervical dilation
Measure: Mean (Standard Deviation); unit: number of side effects out of seven
Units Other Than Participants: side effects
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 7 | 3
Number analyzed (side effects) | 7 | 7
number of side effects out of seven | 0.6 (0.1) | 0.6 (0.3)

3. Secondary Outcome: Dilation Time in Minutes
Description: Time from beginning of cervical dilation to completion of cervical dilation.
Time Frame: At time of procedure.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 7 | 3
minutes | 1.9 (1.1) | 1.4 (.4)

4. Secondary Outcome: Maximum Dilator Size
Description: The largest cervical dilator that could be passed through the internal cervical os.
Time Frame: At time of procedure.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 7 | 3
millimeters | 10.3 (4.8) | 6 (0)

5. Secondary Outcome: Number of Complications
Description: Count of complications at time of surgery.
Time Frame: At time of procedure.
Measure: Mean (Standard Deviation); unit: complications
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 7 | 3
complications | 0.1 (0.4) | 0 (0)

6. Secondary Outcome: Resistance Score
Description: Ease of Dilation Per Surgeon on a numeric scale of 1(easier than normal) to 5 (more difficult than normal) with 3 being "normal."
Time Frame: At time of procedure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 7 | 3
units on a scale | 2.9 (2) | 2.7 (0.6)

ADVERSE EVENTS:
Arm/Group | Misoprostol Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/3
Other Adverse Events (participants affected / at risk) | 0/8 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No